CLINICAL TRIAL: NCT00724152
Title: Cognitive-behavioral Therapy for Tinnitus
Brief Title: Cognitive Behavioral Therapy (CBT) for Tinnitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C6324-P
Record Dates: First submitted 2008-07-23; First posted 2008-07-29 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Tinnitus
Keywords: coping skills; psychology; audiology; veterans; tinnitus; adult; intervention studies; tinnitus, noise induced; noise; auditory perception
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1/Cognitive Behavioral Therapy (Experimental): Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, etc.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Arm 2/Tinnitus Education (Active Comparator): Participants randomly assigned to this group received six weeks of tinnitus education. Tinnitus education and skills related to attention control, sleep hygiene and relaxation training such as imagery techniques were provided. Tinnitus education included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources.
  Interventions: Behavioral: Tinnitus Education
- Arm 3/Standard Care (No Intervention): Participants randomly assigned to this control group received only standard care. Standard care involves audiological measurement and brief education during the standard care appointment.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — A psychotherapeutic approach to tinnitus management which includes tinnitus education
  Other Names: CBT
  Arms: Arm 1/Cognitive Behavioral Therapy
Behavioral: Tinnitus Education — An audiologic rehabilitative approach to tinnitus education.
  Arms: Arm 2/Tinnitus Education

SUMMARY:
This study examined how useful it is to teach veterans coping skills for dealing with tinnitus, also called ringing in the ears. A psychological intervention, cognitive-behavioral therapy, was used to teach coping skills even though tinnitus is not a psychological disorder. Participants in Period 1 of the study were assigned to one of two groups for the duration of the study and were blinded to their group assignment until the end of the study. One group received education about tinnitus. The other group received education about tinnitus plus additional ways to cope with problems associated with tinnitus such as sleep disturbance and frustration. Participants were selected to participate if their tinnitus was severe and they had been exposed to loud sound. Participants attended up to six weekly group meetings. It was predicted that participants who were randomly assigned to the cognitive behavioral therapy group would report a greater reduction in tinnitus severity than education controls. During Period 2 of the study, a third "standard care" arm was added. Baseline and outcome data of the 4 participants who completed the study after this third arm was added to the study design are not reported.

DETAILED DESCRIPTION:
The objectives of this study were to (1) develop a novel, integrative, psychological intervention, specifically cognitive-behavioral therapy (CBT), for the treatment of tinnitus among veterans who have past exposure to loud noise, and (2) accrue preliminary data examining the efficacy of the approach relative to standard care with education (ED) control conditions. Tinnitus was the most common service-connected disability among veterans 2006-2012. Interventions for tinnitus are few and no cure exists. This pilot study examined the feasibility and efficacy of providing individualized (CBT) for veterans with bothersome tinnitus. Twenty-five veterans were recruited and randomly selected to one of two conditions during Period One of the study; the treatment condition (CBT) or (ED) control. A CBT manual and an ED manual were developed for this study. Subjects were be eligible for the study if their tinnitus was likely caused by noise exposure, their tinnitus was chronic (> 6 months), tinnitus was a major health concern for them, and participants were able to commit to a 6-week course of treatment at the West Haven location of VACHS. Subjects were veterans blinded to the treatment group to which they are assigned if ED or CBT. The THI served as the primary outcome measure and the TRQ served as the secondary outcome measure pre- and post-treatment follow-up. Results of this pilot project were used to inform the design and methods of future rigorous randomized controlled clinical trials of CBT for tinnitus following its incorporation into the Progressive Tinnitus Management (PTM) protocol. Baseline and outcome data of the 4 participants who completed the study after this third arm was added to the study design are not reported as this third arm essentially modified the design such that a new study began but was not completed.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were veterans who are currently receiving care at VACHS.
* Subjects were interested in participating in the study and had moderate to severe, chronic (>6 months) tinnitus.

  * Following a brief assessment of tinnitus severity by the project coordinator, the research otologist and research audiologist conducted tinnitus and audiological evaluations to determine subject eligibility.
  * The most likely etiology of subjects' tinnitus was noise exposure to and all eligible participants reported having been exposed to loud sound some time in their lives.
* Subjects indicated that they were motivated to comply with treatment and able to commit to a 6-week course of treatment, follow-up, and study participation by continuing to reside nearby.
* Subjects had stable, permanent housing and transportation means for follow-up appointments.
* Tinnitus was a significant health concern for all subjects.
* Women and minorities were recruited.

Exclusion Criteria:

* Subjects responded to five assessment measures to determine exclusion from the study.

  * Tinnitus-Impact Screening Interview (TISI): Those who scored 4 or lower were excluded from the study.
  * Semi-Structured Clinical Interview for Tinnitus: The exclusionary criteria described below were assessed using this measure.
  * Structured Clinical Interview for Diagnosis, abbreviated - Interview/Non-patient (SCIDa-I/NP): If there was any indication of psychosis on this measure, the subject was excluded from the study.
  * Tinnitus Handicap Inventory (THI): Subjects with scores of 19 or lower were excluded.
  * Tinnitus Reaction Questionnaire (TRQ): Subjects who scored 16 or lower on this measure were excluded from the study.
* Subjects who were undergoing litigation or legal matters related to auditory disorders were excluded from the study.
* Subjects must never had previously received psychological treatment for their tinnitus.
* Subjects with otherwise treatable tinnitus were excluded.
* Subjects who had a history of psychotic disorders or dementia were excluded.
* These psychotic symptoms constituted exclusion from the study:

  * delusions of reference
  * persecutory delusions
  * religious delusions
  * grandiose delusions
  * somatic delusions
  * delusional guilt
  * poverty or nihilism
  * delusions of jealousy
  * delusions of mind reading
  * delusions of being controlled
  * delusions of thought-broadcasting
  * auditory hallucinations
  * visual hallucinations
  * tactile hallucinations
  * gustatory and olfactory hallucinations
* Subjects who report having a recent (within 3-month) history of alcohol or drug abuse or dependence other than tobacco or caffeine were excluded.
* Subjects who presented with sudden or fluctuating hearing loss were excluded.
* Subjects with tinnitus associated with otologic disease (e.g., Meniere's Disease) or other co-occurring diseases affecting vestibular dysfunction were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Kerns, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1/Cognitive Behavioral Therapy: Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources.
Period: Two-arm Study Period
Arm/Group | Arm 1/Cognitive Behavioral Therapy | Arm 2/Tinnitus Education | Arm 3/Standard Care
Started | 14 | 11 | 0 (Standard Care arm was added later (Period 2))
Completed | 11 | 9 | 0
Not Completed | 3 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0
Period: Three-arm Study Period (+Standard Care)
Arm/Group | Arm 1/Cognitive Behavioral Therapy | Arm 2/Tinnitus Education | Arm 3/Standard Care
Started | 4 | 2 | 2 (3-group randomization began)
Completed | 3 | 0 | 1
Not Completed | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Period 1 and Period 2
Groups:
- Period 1: Arm 1/Cognitive Behavioral Therapy: Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 2 grp randomize.
- Period 1: Arm 2/Tinnitus Education: Participants randomly assigned to this group received six weeks of tinnitus education. Tinnitus education and skills related to attention control, sleep hygiene and relaxation training such as imagery techniques were provided. Tinnitus education included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 2 group randomization.
- Period 2: Arm 1/Cognitive Behavioral Therapy: Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 3 grp randomize.
- Period 2: Arm 2/Tinnitus Education: Participants randomly assigned to this group received six weeks of tinnitus education. Tinnitus education and skills related to attention control, sleep hygiene and relaxation training such as imagery techniques were provided. Tinnitus education included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 3 group randomization.
- Period 2: Arm 3/Standard Care: Participants randomly assigned to this control group received only standard care. Standard care involves audiological measurement and brief education during the standard care appointment. 3 group randomization.
- Total: Total of all reporting groups
Arm/Group | Period 1: Arm 1/Cognitive Behavioral Therapy | Period 1: Arm 2/Tinnitus Education | Period 2: Arm 1/Cognitive Behavioral Therapy | Period 2: Arm 2/Tinnitus Education | Period 2: Arm 3/Standard Care | Total
Number analyzed (Participants) | 11 | 9 | 3 | 0 | 1 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.6) | 66.4 (9.5) | 63 (19.5) |  | 60 (0) | 64 (9.7)
Gender [Number; unit: participants]
  Female | 0 | 0 | 0 |  | 0 | 0
  Male | 11 | 9 | 3 |  | 1 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 | 7 | 3 |  | 1 | 19
  African American | 2 | 1 | 0 |  | 0 | 3
  Latino | 0 | 1 | 0 |  | 0 | 1
  Mixed | 1 | 0 | 0 |  | 0 | 1
Tinnitus Handicap Inventory [Mean (Standard Deviation); unit: units on a scale] — The THI score ranges from 0 to 100, with 100 indicating the most severe tinnitus and 0 is the least severe tinnitus.
  units on a scale | 44.1 (20.2) | 55.1 (13.9) | 40.7 (19.6) |  | 30.0 (0) | 49.1 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Handicap Inventory (THI)
Description: Most widely used measure of tinnitus distress available during study period. The THI was created using the Tinnitus Handicap Questionnaire and the Tinnitus Questionnaire as well as the Beck Depression Inventory and Modified Somatic Perception Questionnaire. Its construct validity was also assessed using patients' responses on symptom rating scales and auditory tests of pitch and loudness. The THI score ranges from 0 to 100, with 100 indicating the most severe tinnitus and 0 is the least severe tinnitus. The authors of the THI have designated levels of severity, with scores of 16 and below falling into the "no handicap" range. This measure has strong internal consistency reliability (Cronbach's alpha = .93) and test-retest validity for the total score (r = .92). Significant improvement in tinnitus handicap can be observed with a 20-point change in total score.
Time Frame: pre-treatment (session 1) to post-treatment (session 6; approximately 6 weeks after session 1)
Population: Period 1 and Period 2
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Groups:
- Period 1: Arm 1/Cognitive Behavioral Therapy: Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 2 grp random.
- Period 2: Arm 1/Cognitive Behavioral Therapy: Participants randomly assigned to this experimental group received six weeks of tinnitus education plus cognitive behavioral therapy. Cognitive behavioral therapy for tinnitus participants addressed cognitive and behavioral skills targeting the management of tinnitus and the negative impacts of tinnitus. Long-term self-efficacy and self-sufficiency were emphasized. The major components of CBT for tinnitus included identification of individual responses and beliefs about tinnitus and hearing loss, re-conceptualization of the tinnitus experience as one in which the patient has personal control, presentation of skills to modify cognitions and change behaviors, and reinforcement of skills via goals setting, homework and activities. Skills related to attention control, sleep hygiene, relaxation training are provided. Tinnitus education also included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. 3 grp random.
Arm/Group | Period 1: Arm 1/Cognitive Behavioral Therapy | Period 1: Arm 2/Tinnitus Education | Period 2: Arm 1/Cognitive Behavioral Therapy | Period 2: Arm 2/Tinnitus Education | Period 2: Arm 3/Standard Care
Number analyzed (Participants) | 11 | 9 | 3 | 0 | 1
units on a scale of 0-100 | 37.9 (16.9) | 45.1 (20.0) | 42.67 (23.2) |  | 26.0 (0)
Statistical Analysis 1: Comparison: Period 1: Arm 1/Cognitive Behavioral Therapy vs Period 1: Arm 2/Tinnitus Education; Null hypothesis: The Cognitive Behavioral Therapy group would not demonstrate decreased distress at post-treatment as compared to the Tinnitus Education group on the primary outcome measure (THI) between pre-treatment and post-treatment; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Tinnitus Reaction Questionnaire (TRQ)
Description: This is another commonly used measure of tinnitus distress in research. The TRQ is a global measure of tinnitus distress and was developed using correlations with clinician and self-report ratings of symptom categories. Scores on this measure range from 0 to 104 with higher scores indicating more distress. This measure has a high internal consistency reliability (Cronbach's alpha = .96) and test-retest validity for the total score (r = .88). Scores of 17 points or higher on this measure will indicate tinnitus severity is such that the patient is significantly disturbed by tinnitus. This is based on the use of the TRQ as a pre-test measure in measuring outcome of a controlled trial of CBT for tinnitus in an elderly sample. That study sample had an average TRQ score of 16.9 prior to treatment.
Time Frame: pre-treatment (session 1) to post-treatment (session 6; approximately 6 weeks later)
Population: Period 1 and Period 2
Measure: Mean (Standard Deviation); unit: units on a scale ranging 0-104
Arm/Group | Period 1: Arm 1/Cognitive Behavioral Therapy | Period 1: Arm 2/Tinnitus Education | Period 2: Arm 1/Cognitive Behavioral Therapy | Period 2: Arm 2/Tinnitus Education | Period 2: Arm 3/Standard Care
Number analyzed (Participants) | 11 | 9 | 3 | 0 | 1
units on a scale ranging 0-104 | 24.3 (21.6) | 31.2 (16.7) | 29.3 (11.4) |  | 15.0 (0)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Arm 2/Tinnitus Education: Participants randomly assigned to this group received six weeks of tinnitus education.
  Tinnitus education and skills related to attention control, sleep hygiene and relaxation training such as imagery techniques were provided. Tinnitus education included causes, treatments, current research, epidemiological information, basic anatomy of the ear and brain, and support resources. Participants randomly assigned to this control group received only standard care. Standard care involves audiological measurement and brief education during the standard care appointment.
Arm/Group | Arm 1/Cognitive Behavioral Therapy | Arm 2/Tinnitus Education | Arm 3/Standard Care
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/13 | 0/2
Other Adverse Events (participants affected / at risk) | 0/18 | 0/13 | 0/2

LIMITATIONS AND CAVEATS:
During Period 2 only two participants (one completer) were randomized to "standard care" and only four participants (3 completers) were randomized "Cognitive Behavioral Therapy."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No